CLINICAL TRIAL: NCT04806802
Title: 7 Day Trial of APIOC Sphere and APIOC Astigmatism
Brief Title: APIOC Sphere and APIOC Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lentechs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEN102
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Myopia; Hyperopia; Astigmatism
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- APIOC Sphere or Astigmatism (Experimental): Single Vision Spherical or Toric Contact Lens
  Interventions: Device: APIOC Sphere and APIOC Astigmatism

INTERVENTIONS:
Device: APIOC Sphere and APIOC Astigmatism — Single Vision Contact Lenses

SUMMARY:
Vision and comfort, both objective and subjective, will be assessed for single vision contact lens wearers for either the APIOC™ Sphere or the APIOC™ Astigmatism contact lenses.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must provide written informed consent.
2. The subject must appear willing and able to adhere to the instructions set forth in this protocol.
3. At least 18 years of age and no more than 35 years of age.
4. ≤ 4.00 D (diopters) of corneal astigmatism.
5. ≤ 2.50 D of refractive astigmatism.
6. Refractive error range +4.00 DS to -6.00 DS (diopters sphere)
7. Flat and steep keratometry readings within 40 to 48 D.
8. Clear, healthy corneas with no irregular astigmatism.
9. Normal, healthy conjunctiva in both eyes.
10. Free of active ocular disease. Refractive error is permitted.
11. Be a current or former (within the last 12 months) contact lens wearer.
12. Best-corrected near and distance visual acuity better than or equal to 20/25.

Exclusion Criteria:

1. Irregular corneal astigmatism.
2. Presbyopia
3. Corneal scarring unless off line-of-site and well healed.
4. Pinguecula, pterygium, or other conjunctival thickness abnormalities that would interfere with soft contact lens wear.
5. Recent use of any ocular pharmaceutical treatments, including daily artificial tears, in the two weeks prior to the examination. Use of artificial tears less than 3 drops per week is permitted.
6. Systemic disease that would interfere with contact lens wear.
7. Currently pregnant or lactating (by self-report).
8. History of strabismus or eye movement disorder, including exophoria at near that is 4 D or greater than at far, and a receded near point of convergence break that is 6 cm or greater.
9. Active allergies that may inhibit contact lens wear.
10. Upper eyelid margin at or above the superior limbus.
11. History of ocular or lid surgery.
12. Immediate family members or significant others of doctors or staff at the clinical site.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | Day 7
  High and Low Contrast LogMAR, Distance
Subjective Vision Quality | Day 7
  Visual analogue scale
Comfort | Day 7
  Visual analogue scale

SECONDARY OUTCOMES:
Subjective comfort | Day 7
  Compared to habitual lenses
Subjective vision | Day 7
  Compared to habitual lenses

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Complete Family Vision Care, San Diego, California
  - Eola Eyes, Orlando, Florida
  - Gaddie Eye Centers, Lexington, Kentucky
  - Miamisburg Vision Care, Miamisburg, Ohio
  - Vision Professionals, New Albany, Ohio
  - Eyecare Professionals of Powell, Powell, Ohio

IPD SHARING:
Plan to Share IPD: No
No sharing of data is planned.